CLINICAL TRIAL: NCT07225829
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Proof of Concept Trial to Investigate the Efficacy and Safety of Intra-articular 4P004 in Subjects With Knee Synovitis and Osteoarthritis
Brief Title: A Trial to Investigate the Safety and Efficacy of Intra-articular 4P004 Injection in Subjects With Knee Synovitis and Osteoarthritis
Acronym: INFLAM MOTION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 4Moving Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4MB-4P004-P-INFLAM; 2024-518916-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-24; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis; Synovitis of Knee
Keywords: OA; Knee OA; Liraglutide; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Liraglutide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A total of one hundred and twenty-nine (129) participants will be randomized in the trial, and enrolled in two arms. Participants in the active arm will receive one intra-articular (IA) injection of 4P004 (2mL), while the placebo arm will receive 2mL of NaCl 0.9%. Randomization ratio will be 2:1 (4P004:Placebo).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4P004 (2mL) (Experimental): One IA injection in the knee of 4P004 (2mL) on the day of randomization
  Interventions: Drug: 4P004
- Placebo (NaCl 0.9% 2mL) (Placebo Comparator): One IA injection in the knee of Placebo (NaCl 0.9% 2mL) on the day of randomization
  Interventions: Drug: Placebo (NaCl 0.9%)

INTERVENTIONS:
Drug: 4P004 — Single intra-articular injection in the knee joint
  Other Names: Liraglutide
  Arms: 4P004 (2mL)
Drug: Placebo (NaCl 0.9%) — Single intra-articular injection in the knee joint
  Arms: Placebo (NaCl 0.9% 2mL)

SUMMARY:
This phase 2a trial is an international, multicenter, randomized, double-blind, placebo-controlled trial to investigate the efficacy and safety of one single intra-articular (IA) injection of 4P004 or placebo in:

* patients between 40 and 80 years of age,
* with synovitis and grade 2 to 4 osteoarthritis (OA) of the knee according to Kellgren and Lawrence (KL) classification.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have the capacity to give informed consent and who are willing to comply with all trial related procedures and assessments.
* Participants between 40 and 80 years of age.
* Female participant of childbearing potential (defined as any woman unless postmenopausal for at least one year or surgically sterile) must use highly effective methods of contraception as defined in the protocol. Highly effective contraceptive measures must be continued throughout the trial until the final visit.
* Bodyweight > 40 kg.
* Body mass index (BMI) ≥ 18.5 and ≤ 35.
* Ambulatory (single assistive devices such as canes allowed).
* Widespread Pain Index (WPI) ≤ 4.
* Pain NRS (0-10) < 4 in the contralateral knee.
* History of OA-related pain of the TK for at least 6 months.
* Moderate to severe pain of the TK the majority of days during the last 3 months as per participant's judgement.
* Moderate to severe pain of the TK on the WOMAC Pain subscale prior to the Randomization visit (V2) complying with: a) Complete WOMAC Pain diary for at least 7 of the last 10 days prior to V2 (including V2/D1 rating which is mandatory), and b) Diary reported WOMAC Pain between 5 and 9 for at least 7 of the last 10 days.
* History of insufficient pain relief, intolerance, or contraindication to NSAIDs, and at least a history of insufficient pain relief from at least one of the following therapies: a) Acetaminophen/paracetamol, b) Opioids including tramadol, or c) Corticosteroids, hyaluronate IA injections (efficacy less than 3 months according to the patient).
* KL grade 2 to 4 on the Schuss radiograph.
* Predominant femorotibial OA based on the OA Research Society International. (OARSI) Atlas reading (Altman & Gold, 2007).
* Presence of synovitis in the TK assessed locally using PDUS, and synovial thickness of ≥ 5 mm evaluated through a longitudinal view of the suprapatellar pouch and axial views of the medial and lateral patellofemoral pouches.
* Negative urine drug screen (performed locally): amphetamines, barbiturates, cocaine.
* CE-MRI Central reading to confirm synovitis with a synovial Semi-Quantitative (SQ) ≥ 9 or a SQ score ≥7 with at least one site with a score ≥ 2.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the TK (varus > 10°, valgus > 10°) by radiography.
* Secondary OA such as joint dysplasia, aseptic osteonecrosis, joint infection, acromegaly, Paget disease, hemochromatosis, joint crystal disease or any inflammatory joint disease.
* Any known active infections including skin infections at the site injection or increased predisposition for the development of infections.
* Any partial knee replacement of the TK.
* Acute fracture or IA trauma to the TK within 12 months prior to the screening visit.
* Major knee surgery performed within the previous 12 months or planned during the trial.
* Arthroscopy of the TK within 6 months prior to the screening visit.
* Presence of any painful conditions that could confound accurate assessment of pain from OA in the TK, such as fibromyalgia, peripheral neuropathy or vascular insufficiency.
* Treatment with systemic corticosteroids (other than IA) at a dose greater than 10 mg prednisone or the equivalent per day for more than 7 days within 4 weeks prior to the screening visit.
* Treatment of the TK with any IA injection (including corticosteroids, hyaluronic acid derivatives, Platelet Rich Plasma….) within 24 weeks prior to the screening visit.
* Any treatment with glucosamine, chondroitin sulfate, or other nutraceuticals with potential activity on OA within the previous 3 months prior to the screening visit.
* Treatment with duloxetine for OA (allowed if given for depressive disorders at stable dose since at least 3 months before V1).
* Any significant psychiatric illness unless well controlled since at least 6 months.
* Current treatment with combination of insulin and liraglutide (Xultophy®) or with GLP-1 agonist administered once a week (semaglutide, dulaglutide).
* High-risk of bleeding.
* Congestive Heart Failure stage III or IV in the New York Heart Association classification.
* History or current diagnosis of electrocardiogram ECG abnormalities indicating significant safety risk (such as ischemia, significant cardiac arrhythmias).
* Glycemia < 4.4 mmol/L (or 80 mg/dL) at screening.
* Clinically significant abnormal laboratory test at screening, in particular: haemoglobin <10 g/dL, white blood cell <3000/µL (3.0 Giga/L), absolute neutrophil count <1000/µL (1.0 Giga/L), platelets count <100,000/µL (100 Giga/L), alanine aminotransferase or aspartate aminotransferase >2.5 upper limit of normal (ULN), total bilirubin >1.5 ULN, lipasemia >1 ULN.
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2, using Chronic Kidney Disease - EPIdemiology (CKD EPI) 2021 Formula.
* Any other abnormal laboratory results that the Investigator believes should preclude the subject's participation in the trial.
* History of hypersensitivity to IMP or excipients (liraglutide or disodium phosphate dihydrate, propylene glycol, phenol).
* Any contraindication for MRI (cardiac pacemaker, deep brain stimulators, intraocular metal, cerebral aneurysm clips, recent stents, cochlear implants, neurostimulators and implantable pumps) or inability to undergo MRI (e.g., body size, leg not fitting in the coil, claustrophobia).
* History of hypersensitivity reactions to a gadolinium-based contrast agent.
* Any CE-MRI Central reading additional diagnoses: posterior meniscal root tears, subchondral insufficiency fractures, osteonecrosis, malignant bone marrow infiltration, solid tumours, and traumatic fracture or bone bruise using ROAMES (Roemer et al., 2020).
* Previous participation in clinical research with a disease-modifying OA drug during the last 2 years.
* Participation in an interventional clinical research trial within 3 months before screening.
* Participants who, in the investigator's judgement, are at risk of falling.
* Participants with a history, or current diagnosis, of pancreatitis, thyroid cancer (including medullary thyroid carcinoma), multiple endocrine neoplasia type-2 (MEN2), diabetic ketoacidosis, type-1 diabetes mellitus (T1DM), inflammatory bowel disease, or diabetic gastroparesis.
* Participants currently, or within the last 10 days, taking any anticoagulant treatment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline at Week 4 in the weekly average of Target Knee (TK) daily pain intensity using the WOMAC (Western Ontario and McMaster Universities Arthritis Index) Pain subscore | Baseline and Week 4
  The WOMAC is a questionnaire widely used in the evaluation of knee osteoarthritis. It contains 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items). Scores are calculated for each subscale and summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Change from Baseline at Week 2, Week 6, Week 8, Week 10 and Week 12 in the weekly average of TK (Target Knee) daily pain intensity using the WOMAC (Western Ontario and McMaster Universities Arthritis Index) Pain subscore | Baseline, Week 2, Week 6, Week 8, Week 10 and Week 12
  The WOMAC is a questionnaire widely used in the evaluation of knee osteoarthritis. It contains 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items). Scores are calculated for each subscale and summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Change from Baseline at Week 2, Week 4, Week 8 and Week 12 in the NRS (Numeric Rating Scale) pain (scale 0-10) in a nominated pain aggravating activity | Baseline, Week 2, Week 4, Week 8 and Week 12
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time, using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
Change from Baseline at Week 2, Week 4, Week 8 and Week 12 in WOMAC (Western Ontario and McMaster Universities Arthritis Index) subscores and total score | Baseline, Week 2, Week 4, Week 8 and Week 12
  The WOMAC is a questionnaire widely used in the evaluation of knee osteoarthritis. It contains 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items). Scores are calculated for each subscale and summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Change from Baseline at Week 2, Week 4, Week 8 and Week 12 in the Patient Global Assessment of Osteoarthritis (PGA-OA) | Baseline, Week 2, Week 4, Week 8 and Week 12
  The PGA-OA is a 1-item questionnaire designed to assess the participant's impression of disease severity adapted from Guy et al., 1976, to the specific disease as a Patient-reported Outcome measurement "Considering all the ways your knee osteoarthritis affects you, how are you doing these last seven days ?".
  PGA-OA is measured on a 5-point Likert scale, with higher scores indicating worse symptoms (1= "very good" to 5 = "very poor").
Percentage (%) of OMERACT-OARSI Responders at Week 2, Week 4, Week 8 and Week 12 | Week 2, Week 4, Week 8 and Week 12
Incidence and severity of TEAEs (Treatment-Emergent Adverse Events) during the trial | From randomization to end of trial, up to 12 weeks
Absolute changes from Baseline in clinical laboratory assessment - hematology parameter: total blood cells count (in cell/L) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in clinical laboratory assessments - hematology parameter: hemoglobin (in g/L) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in clinical laboratory assessment - blood chemistry: AST (in U/L) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in clinical laboratory assessment - blood chemistry: ALT (in U/L) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in clinical laboratory assessment - blood chemistry: lipase (in U/L) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in clinical laboratory assessment - blood chemistry: fasting glycemia (in mmol/L) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in clinical laboratory assessment - blood chemistry: total bilirubin (in umol/L) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in Vital signs: systolic and diastolic blood pressure (BP) | From randomization to end of trial (up to 12 weeks)
Absolute changes from Baseline in Vital signs: pulse rate | From randomization to end of trial (up to 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Berenbaum, MD, PhD, Study Chair — 4
Locations (21):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Skylight Health Research Burlington, Burlington, Massachusetts
- Canada (3):
  - Durham Bone and Joint Specialists, Ajax
  - SJHC London Rheumatology Centre, London
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc, Québec
- Denmark (2):
  - Parker Institute Bispebjerg, Frederiksberg Hospital, Frederiksberg
  - Sanos Clinic Herlev, Herlev
- France (5):
  - CHU Montpellier, Montpellier
  - ChU de Nice, Nice
  - Hôpital Cochin, Paris
  - Hôpital Lariboisière, Paris
  - Centre Hospitalier Universitaire CHU de Reims - Hopital Maison Blanche, Reims
- Poland (3):
  - Care Access Kraków, Krakow
  - Centrum Medyczne Reuma Park, Warsaw
  - MICS Centrum Medyczne Warszawa, Warsaw
- Spain (6):
  - Complejo Hospitalario Universitario de A Coruna - Hospital Universitario de A Coruna, A Coruña
  - HLA Clínica Vistahermosa, Alicante
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Sabadell
  - Hospital Universitario Marques de Valdecilla, Santander
  - Clinica Nuestra Senora de la Esperanza, Santiago de Compostela
  - Hospital Quirónsalud Sagrado Corazón, Seville

IPD SHARING:
Plan to Share IPD: Undecided